CLINICAL TRIAL: NCT04985331
Title: Randomized Controlled Trial of a Digital Therapeutic Versus Psychoeducation for the Management of Mild to Moderate Depression in Adolescents
Brief Title: Digital Therapeutic vs Psychoeducation for Management of Mild to Moderate Depression in Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Woebot Health (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: W-GenZD-002
Record Dates: First submitted 2021-07-08; First posted 2021-08-02 (Actual); Last update posted 2022-01-05 (Actual); Status verified 2022-01

CONDITIONS: Depression, Teen
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- W-GenZD (Experimental): W-GenZD is powered by natural language processing and machine learning techniques, the brief, self-guided intervention draws from cognitive behavioral therapy (CBT), interpersonal psychotherapy (IPT-A) and some elements of dialectical behavior therapy (DBT), depending on the presenting situation, to help the adolescent develop emotion regulation skills in the context of their everyday life. In this way, the mobile medical application is designed to be targeted, relevant, tailored, and integrated into the lived experience of adolescents, capable of delivering the appropriate technique for the problem at hand, at the time of need.
  Interventions: Device: W-GenZD
- Psychoeducation Control (No Intervention): The control for this study is the scheduled delivery of digital psychoeducational files (PDFs). The PDFs were selected to provide information on depression, anxiety and stress, as well as outline common coping skills.

INTERVENTIONS:
Device: W-GenZD — W-GenZD is a program that delivers evidence based therapy for the symptoms of mild-moderate depression and anxiety in adolescents in brief "conversations" with a fully automated relational agent.
  Arms: W-GenZD

SUMMARY:
The purpose of the present randomized controlled study is to investigate if there is a difference in depression symptoms at 4-weeks among adolescents ages 16-17 years assigned to W-GenZD, a digital therapeutic, as compared to a psychoeducational control group.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents aged 16-17 years old
* Experiencing mild-moderate depression as indicated by a PHQ-8 score between 5-19, inclusive, assessed at screening/baseline
* Has regular access to a smartphone (Android or iOS smartphone with a recent supported operating system) with reliable WiFi access or sufficient data to engage with assigned study arm for the duration of the study
* Available and committed to engage with the program and complete assessments for an 8-week duration
* Able to read and write in English
* U.S. resident
* Regular, stable dose of antidepressant medications for (e.g. escitalopram/Lexapro, fluoxetine/ Prozac) for at least 60 days at screening with no plans to change medication/dose throughout the study
* If currently receiving psychotherapy, then must be in therapy for at least 4 weeks at screening with no changes planned for the duration of the study
* Participants must be able to understand and willing to provide informed assent and to comply with all study procedures and restrictions

Exclusion Criteria:

* Lifetime diagnosis of a psychotic disorder, including schizophrenia and schizoaffective disorder
* Lifetime diagnosis of bipolar disorder
* Lifetime diagnosis of autistic spectrum disorder or pervasive developmental disorder (e.g. autism, Asperger syndrome, Rett's syndrome, or pervasive developmental disorder not otherwise specified)
* Suicidal attempt or ideation with a plan and intent to harm oneself during the last 12 months
* History of (a) drug and/or alcohol abuse within the past 12 months (determined by self-report)
* Current use of benzodiazepines (e.g. lorazepam, clonazepam, alprazolam, diazepam, triazolam) or certain sleep aids (zolpidem, eszopiclone, zaleplon)
* Previous Woebot Application use

Ages: 16 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 246 (Actual)
Dates: Start 2021-08-02 (Actual); Primary Completion 2021-12-16 (Actual); Study Completion 2022-01-04 (Actual)

PRIMARY OUTCOMES:
Patient Health Questionnaire (PHQ-8) | Change from Baseline to Mid-Treatment at 2 weeks; Change from Baseline to Post-treatment at 4 weeks; Change from Baseline to 1-Month Follow-up at 8 weeks
  Measure of depression severity. Total score between 0-27, where higher scores indicate greater levels of depression.

SECONDARY OUTCOMES:
Generalized Anxiety Disorder (GAD-7) | Change from Baseline to Mid-Treatment at 2 weeks; Change from Baseline to Post-treatment at 4 weeks; Change from Baseline to 1-Month Follow-up at 8 weeks
  Measure of anxiety. Total score between 0-21, where higher scores indicate greater levels of anxiety.
Working Alliance Inventory (WAI-SR) | Difference between mid-treatment at 3 days weeks within treatment and post-treatment at 4 weeks
  Therapeutic alliance that assesses three key aspects of the therapeutic alliance: (a) agreement on the tasks of therapy, (b) agreement on the goals of therapy and (c) development of an affective bond. Scores range from 5-20, with higher scores indicating greater alliance.
Mental Health Self-Efficacy Scale (MHSE) | Change from Baseline to Post-treatment at 4 weeks; Change from Baseline to 1-Month Follow-up at 8 weeks
  Assesses confidence in managing stress, depression, and anxiety. Range is 10 to 60, with higher scores indicating more self-efficacy.
Client Satisfaction Questionnaire (CSQ) | Post-treatment (8 weeks from baseline)
  Range from 8 to 32, with higher values indicating higher satisfaction
Usage Rating Profile Intervention (URPI) | Post-treatment (8 weeks from baseline)
  Measurement of feasibility and acceptability. Scores range from 6-36, with higher scores indicating greater feasibility and acceptability.
Number of active application days | Post-treatment (8 weeks from baseline)
  Application engagement in the total number of active days using the application will be collected during the study to provide quantitative data regarding application utilization.
Number of application messages sent per week | Post-treatment (8 weeks from baseline)
  Application engagement in the number of messages sent each week within the application will be collected during the study to provide quantitative data regarding application utilization.
Satisfaction ratings of psychoeducational materials | Post-treatment (8 weeks from baseline)
  Satisfaction metrics in the total number of 'Thumbs up' (likes) or 'Thumbs down' (dislikes) will be collected during the study to provide quantitative data regarding satisfaction with program content.
Mood change ratings after CBT skill application | Post-treatment (8 weeks from baseline)
  Satisfaction metrics in the total number of mood change ratings of 'same', 'better', or 'worse, after learning a CBT skill application will be collected during the study to provide quantitative data regarding satisfaction with content.

CONTACTS AND LOCATIONS:
Locations (1):
- Woebot Health, San Francisco, California, United States